CLINICAL TRIAL: NCT02672722
Title: Assessment of the Changes in Cortical and Medullary Renal Blood Flow During Exercise in Healthy Subjects Using Contrast Enhanced Ultrasound
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Kambiz Kalantarinia, MD, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18220
Record Dates: First submitted 2016-01-25; First posted 2016-02-03 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Healthy; Physiology
Keywords: This term was found doing the MeSH search and is the only thing that fits since we will be working with healthy subjects with no conditions.
MeSH Terms: interventions — perflutren; Microbubbles; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy Test Subjects (Experimental): We will be using the drug Definity that is an approved medication for cardiac contrast enhanced ultrasound to measure the changes in kidney blood flow with exercise in healthy subjects.
  Interventions: Drug: Definity; Other: Exercise; Other: Kidney Ultrasound

INTERVENTIONS:
Drug: Definity — During kidney ultrasound, Definity microbubbles will be injected into the vein to see how blood flows through the kidneys
  Other Names: ultrasound contrast agent or microbubbles
Other: Exercise
  Other Names: stationary Bike
Other: Kidney Ultrasound — This done before and after exercise with the help of Definity to see changes in kidney blood flow
  Other Names: Renal Ultrasound examination

SUMMARY:
Renal parenchymal blood flow can be divided in cortical and medullary blood flow. Changes and factors affecting renal medullary blood flow have not been studied in detail previously as investigators/doctors did not have tools to monitor renal medullary blood flow in vivo. Since Trueta first described renal medullary blood flow, multiple attempts have been made to study renal medullary blood flow using invasive methods. Recently renal medullary blood flow measurement using contrast US has emerged as a promising technique that investigators can use to study renal medullary blood flow in vivo. In this study investigators are aiming to study changes in renal parenchymal (cortical and medullary) blood flow with exercise in healthy subject.

DETAILED DESCRIPTION:
This study requires a screening day and two visits on separate days to the Clinical Research Unit (CRU). Three visits total.

Screening Visit:

1. The subjects will undergo detailed history and physical examination.
2. The inclusion and exclusion criteria will be reviewed.
3. The details of the study procedures, potential risks and benefits will be reviewed with each subject and all potential questions will be answered.
4. Subjects' understating of all details of the study components will be ascertained and they will be asked to sign the informed consent form.
5. A copy of the signed informed consent will be placed in study file and another copy will be provided to each subject.
6. The study visit day will be scheduled within 2 weeks of the screening day.
7. All subjects will be asked to arrive on their first study day after an overnight fast. They will be instructed to avoid caffeine and exercise for 24 hours.

Study Day #1 The subjects will arrive in the CRU in the morning. Subjects' understanding of all study related procedures will be assessed and all remaining questions will be answered. The following sequence of procedures will be followed for all enrolled subjects.

1. Physical exam including vital signs (Blood Pressure, Heart Rate, Weight, Height, Respiration Rate, Temperature)
2. Urine pregnancy test for women of child bearing age. If positive, subjects will be excluded.

   Determination of peak oxygen consumption
3. Subjects will complete a continuous VO2 peak bicycle ergometer protocol.

   1. Each subject will start peddling on a stationary bike
   2. The initial power output (PO) will be set at 20 watts
   3. The power output will be increased by 15 watts every 2-minutes until volitional exhaustion.
   4. Metabolic data will be collected during the protocol using standard open-circuit spirometric techniques (Viasys Vmax Encore, Yorba Linda, CA)
   5. Heart rate was assessed electrocardiographically.
   6. VO2 peak will be chosen as the highest VO2 attained during the exercise protocol

On Day 2 of testing

1. Check Vitals (BP, HR, Wt., RR, Temp.)
2. Insert peripheral IV line Baseline renal blood flow measurement using contrast enhanced ultrasonography
3. The Definity vial will be placed at room temperature before being used. It will be activated after shaking the vial using Vialmax® for 45 seconds. It will be used immediately after activation.
4. 0.4 ml of Definity will be mixed in 10 ml of preservative free saline.
5. Infusion of Definity into a peripheral vein will be started at 2 ml/min and titrated for optimal image quality using a minipump (not to exceed 10 ml/min at any time).
6. Baseline contrast ultrasound imaging of right kidney will be performed with low mechanical index (MI) of 0.2.
7. 4 - 5 ultrasound impulses with high MI of 1.0 and duration of 1 second will be used to destruct the microbubbles in the kidney tissue
8. Ultrasound imaging of the kidney with low MI (0.2) will continue immediately after each impulse for several seconds.
9. Infusion of Definity will stop at this point.
10. Vital signs will be monitored every 15 minutes and continuous pulse oximetry will be performed during Definity administration.
11. Vital signs and pulse oximetry will be monitored every 15 minutes until 30 minutes after discontinuation of Definity.
12. A urine dipstick will be performed by the study team 30 minutes after completion of Definity infusion if a sample is available.

    Constant load Exercise protocol
13. Subjects will complete 30 minutes of continuous cycling at the power output associated with 85% of VO2peak from the continuous bicycle ergometer protocol. Metabolic data will be collected as described above.
14. Once metabolic parameter are reached, exercise will be stopped and subject will be asked to lie down on the bed Renal Blood flow measurement following exercise using contrast enhanced ultrasonography
15. Immediately after completion of exercise protocol, steps 5 - 12 under day 2 procedures will be repeated.
16. The study procedures will end at this point.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Adult - 18 to 50 years old
* All ethnicity and genders

Exclusion Criteria:

* Pregnancy or lactation
* Active infection
* Hypertension
* Chronic Medication Use except Multi Vitamin Use and Birth Control Medications
* Known history of a right to left intra-cardiac shunt
* Known history of pulmonary hypertension, including porto-pulmonary hypertension
* History of allergies to Definity®
* History of Liver or Kidney Transplant
* Patient on hemodialysis
* Has received iodinated contrast within 72 hours of admission to study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2017-08 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Change in renal blood flow in exercise as assessed by CEUS | Before and immediately after exercise
  Total, cortical and medullary kidney blood flow will be measured using contrast-enhanced ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Kambiz Kalantarinia, MD, Principal Investigator — University of Virginia, Department of Nephrology
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States